CLINICAL TRIAL: NCT05033782
Title: Impact of the Modifications of Environmental Exposures and Health Care Access During COVID-19 Lockdown on the Risk of Multiple Sclerosis Clinical Relapse or Clinical Worsening
Brief Title: Impact of the Modifications of Environmental Exposures and Health Care Access During COVID-19 Lockdown on Multiple Sclerosis
Acronym: CONFISEP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210935
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; Lockdown; COVID-19; Air pollution; Influenza, Human; Gastroenteritis; Health Services Accessibility
MeSH Terms: conditions — Multiple Sclerosis; COVID-19; Influenza, Human; Gastroenteritis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS patients: This group includes patients living in Ile de France, followed in the neurology department of the Pitié Salpêtrière Hospital in Paris for relapsing-remitting MS.
  Clinical examination will be performed to evaluate the disability (EDSS scale), as part of the care (systematic for all MS consultations)
  - A paper questionnaire is given to the patient during the consultation. The patient will be contacted by telephone within 15 days after the consultation by a health care staff to collect the answers to the questionnaire.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Each included patient will be given a paper questionnaire, with the following questions:
  * Zip code of patient's iterative residences since 2018, as well as the zip code of residence at the time of the 2 confinements
  * Occupational status
  * Occurrence of COVID infection/date needed for hospitalization
  * During the COVID-19 outbreak, did the patient: avoid seeing a doctor, avoid going to health care facilities, stop background treatment for MS. If yes to any of the questions, the reason, date and duration of the cessation will be asked.
  Other sources of data will be used together:
  Clinical data from the OFSEP registry Pollution data from approved air quality monitoring associations Data on the circulation of influenza and gastroenteritis, produced by Santé Publique France

SUMMARY:
Multiple Sclerosis (MS) is a demyelinating auto immune disease of the central nervous system, affecting 2500000 people worldwide. Risk factors for MS severity are not yet well-known , but previous studies highlighted that relapse rate increased during influenzae epidemics, and air pollution could be a risk factor for MS relapses. MS is a neurological chronic disease that requires constant medical treatment and regular rehabilitation care. COVID-19 pandemic and restrictive measures taken to limit contaminations have drastically decreased air pollution and seasonal viral infections exposure, but sanitary crisis also limited care access for MS patients (medical treatment, rehabilitation). Therefore, this particular period offers a unique opportunity to evaluate the impact of air pollution, viral infections, and health care access on the severity of MS.

The main objective is to evaluate the impact of air pollution and seasonal viral infections on the risk of MS relapse, using the year 2020 as a quasi-experimental model. The secondary objective will be to evaluate the impact of health care access limitations on the risk of neurological disability accumulation.

This study will include 1500 MS patients, living in Ile de France, followed in the neurological department of "Pitié-Salpêtrière" Hospital. This is a retrospective observational study nested in OFSEP registry (French Multiple Sclerosis Observatory), which is a prospective cohort of MS patients in France. Air pollution data will come from AIRPARIF, and viral infections data will come from "Santé Publique France".

A better knowledge of the impact of air pollution, viral infections, and health care access on the course of MS will enable to better guide information to patients and public health care decisions.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a common autoimmune disease of the central nervous system. The repetition of relapses and their severity will lead in the long term to the accumulation of disability. The risk factors for relapses are still poorly understood, but it is suspected that air pollution and seasonal viral infections may increase the risk of relapse.

The Sars-Cov-2 virus pandemic has abruptly disrupted the daily environment, to date three lock-down periods have been implemented, in France, to limit the spread of COVID 19, the first was from March 17 to May 11, 2020, the second was less strict from October 30 to December 15, 2020, and the third began April 3, 2021. The reduction in road traffic during the first containment was accompanied in Ile de France by a 30 to 50% decrease in fine particulate matter and nitrogen oxide air pollution compared to the previous year. The confinements and the generalized application of barrier measures have also been associated with a clear decrease in the circulation of seasonal viruses, in particular influenza and viral gastroenteritis viruses, compared to the previous year.

To date, the impact of measures to prevent the spread of the Sars-CoV-2 epidemic on the risk of MS relapse has not been studied. However, these periods offer a unique opportunity to assess, in a quasi-experimental model, the impact of air pollution and viral infections on the risk of MS relapse, in a context where these factors have shown large variations compared to the usual seasonal values observed.

The pandemic has also had a profound impact on the health care system, with the corollary that patients with chronic pathologies have had difficulty accessing care, as hospital structures have had to deal with an unprecedented crisis, resulting in the de-scheduling of non-urgent procedures and great difficulty in accessing in-person consultations. Numerous uncertainties concerning the risk of severe COVID-19 in patients treated with immune-modulators or immune-suppressors have led to the suspension or delay of the initiation of immuno-active treatments to prevent the aggravation of the disease. To date, no study has evaluated the impact of changes in the management of MS patients during this particular period and to assess the impact on the progression of neurological disability.

The primary objective of the study will be to determine the impact of environmental risk factors (air pollution, exposure to seasonal viruses) and health care access on the risk of clinical MS relapse, in the context of the lockdown periods, compared to periods prior to the COVID-19 pandemic.

The secondary objective will be to assess the impact of environmental risk factors (air pollution, exposure to seasonal viruses), on the risk of accumulation of MS disability, in the context of the lockdown periods, compared to periods prior to the COVID-19 pandemic.

This study will include patients followed in the neurology department of the Pitié Salpêtrière Hospital in Paris for relapsing-remitting MS, and will be conducted as bellow:

Inclusion visit:

* Conducted during the patient's usual follow-up (consultation / day hospital).
* Information and collection of non-opposition by the investigating neurologist
* Clinical examination to evaluate the disability (EDSS scale), as part of the care (systematic for all MS consultations)
* A paper questionnaire is given to the patient during the consultation. The patient will be contacted by telephone within 15 days after the consultation by a health care staff to collect the answers to the questionnaire.

Different sources of data will be used together:

1. Clinical data from the OFSEP registry (French Multiple Sclerosis Observatory). OFSEP is a national registry in which neurological clinical data of MS patients are prospectively collected.

   (i) Date of first symptoms of the disease (ii) Date of diagnosis (iii) Date of disease relapses, date of first symptoms of the relapse (iv) Neurological disability score at each neurological assessment as assessed by the EDSS score (v) Nature, date of initiation and discontinuation of treatment and reasons for discontinuation (vi) Comorbidities, infectious and neoplastic complications (vii) Education level
2. Data from the telephone questionnaire:

   (i) Zip code of patient's iterative residences since 2018, as well as zip code of residence at the time of the two confinements (ii) Occupational status (iii) Occurrence of COVID infection/date needed for hospitalization (iv) During the COVID-19 outbreak, did the patient: avoid seeing a doctor, avoid going to health care facilities, stop background treatment for MS. If yes to any of the questions, the change(s) was: decided by the patient, recommended by the treating physician, recommended by the neurologist, other (specify) (v) During the COVID-19 outbreak, did the patient stop his or her rehabilitation care (physical therapy, speech therapy)? If yes, date of cessation, duration, reason for cessation (planned, decided by the patient, recommended by the rehabilitation specialist, recommended by the attending physician, recommended by the neurologist)
3. Pollution data from approved air quality monitoring associations (AASQA): for the Ile de France region, this is AIR PARIF, which collects the daily average exposure to fine particles (PM10, PM2.5), ozone (O3), and nitrogen oxides (NO2) at 37 stations in the different departments of Ile de France. The data from the station closest to each patient's home will be analysed.
4. Data on the circulation of influenza and gastroenteritis, produced by Santé Publique France ("Sentinelles" network, OSCOUR network, National Reference Center for Respiratory Infections Viruses).

ELIGIBILITY:
Inclusion Criteria:

* MS defined by the Mac-Donald 2017 criteria
* Age greater than or equal to 18 years
* Relapsing-remitting form
* Patient residing in Ile de France
* Patient included in the OFSEP registry (French Multiple Sclerosis Observatory) with at least one visit before 2020 and at least one after January 2021

Exclusion Criteria:

* Secondary progressive or primary progressive MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in Ile de France and followed in the neurology department of the Pitié Salpêtrière Hospital in Paris for relapsing-remitting MS.
Sampling Method: Non-Probability Sample
Enrollment: 1209 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Relapse | 01/01/2018 - 01/01/2022
  a neurologic deficit associated with an acute inflammatory demyelinating event that lasts at least 24 hours in the absence of fever and infection

SECONDARY OUTCOMES:
Neurological disability accumulation | 01/01/2018 - 01/01/2022
  increase of EDSS of 1.5 points for EDSS <2, and 1 point for EDSS [2-5.5], and 0.5 point for EDSS >5.5.

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Januel, MD, Principal Investigator — Assistance Publique Hopitaux Paris
Locations (1):
- Neurology Department, Hopital de la Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.